CLINICAL TRIAL: NCT06540144
Title: An Open-label Extension Study to Evaluate Rozanolixizumab in Pediatric Study Participants With Generalized Myasthenia Gravis
Brief Title: An Extension Study Evaluating 6-week Treatment Cycles of Rozanolixizumab in Pediatric Study Participants With Generalized Myasthenia Gravis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0008; 2022-502075-34 (Registry Identifier: EU CTIS); U1111-1286-3581 (Other: WHO universal trial number (UTN))
Record Dates: First submitted 2024-07-22; First posted 2024-08-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Generalized Myasthenia Gravis; gMG; rozanolixizumab; pediatric
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- rozanolixizumab (Experimental): Study participants will receive pre-defined doses of rozanolixizumab. Each treatment cycle in each Treatment Period (TP) consists of 6 subcutaneous (sc) administrations of rozanolixizumab at 1-week intervals. Each Treatment Period will be initiated upon the discretion of the Investigator based on the medical needs of the study-participant.
  Interventions: Drug: rozanolixizumab

INTERVENTIONS:
Drug: rozanolixizumab — rozanolixizumab solution for injection
  Other Names: UCB7665

SUMMARY:
The purpose of the study is to assess the long term safety and tolerability of additional 6-week treatment cycles with rozanolixizumab in pediatric participants with generalized Myasthenia Gravis (gMG) aged ≥2 at the time of the Screening Visit of MG0006.

ELIGIBILITY:
Inclusion Criteria:

Study participant must meet one of the following:

* Study participant completed MG0006 according to the protocol
* Study participant completed the MG0006 Treatment Period and has a worsening of generalized myasthenia gravis (gMG) symptoms in the Observation Period of MG0006

Exclusion Criteria:

* Study participant met any mandatory withdrawal or mandatory permanent investigational medicinal product (IMP) discontinuation criteria in MG0006 or permanently discontinued IMP
* Study participant has a known hypersensitivity to any components of the IMP or other neonatal Fc receptor (FcRn) drugs
* Study participant has any laboratory abnormality that, in the opinion of the Investigator, is clinically significant, has not resolved at Baseline, and could jeopardize or compromise the study participant's ability to participate in this study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-08-17 (Estimated); Study Completion 2027-08-17 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serious Treatment-Emergent Adverse Events (TEAEs) up to the End of Study (EOS) Visit | From Baseline up to the EOS Visit (up to 52 weeks)
  Serious TEAEs are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment and additionally are emergent untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent disability/incapacity
  * Is a congenital anomaly or birth defect
  * Important medical events
Occurrence of TEAEs leading to permanent withdrawal of IMP up to the EOS Visit | From Baseline up to the EOS Visit (up to 52 weeks)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Occurrence of Adverse Event(s) of Special Monitoring (AESM) up to the EOS Visit | From Baseline up to the EOS Visit (up to 52 weeks)
  AESMs are: Severe and/or serious headache, suspected aseptic meningitis, severe Gastrointestinal (GI) disorders, and opportunistic infection.

SECONDARY OUTCOMES:
Percent change in total Immunoglobulin G (IgG) from Baseline to the end of Week 6 of each Treatment Period (TP) | From Baseline to the end of Week 6 of each TP (up to 52 weeks)
  Plasma concentration analyses of total IgG will be done for all study participants on an ongoing basis to the end of Week 6 of each TP.
Absolute change in total IgG from Baseline to the end of Week 6 of each TP | From Baseline to the end of Week 6 of each TP (up to 52 weeks)
  Plasma concentration analyses of total IgG will be done for all study participants on an ongoing basis to the end of Week 6 of each TP.
Change from Baseline in Myasthenia Gravis-Activities of Daily Living (MG ADL) total score at the end of Week 6 of each TP | From Baseline to the end of Week 6 of each TP (up to 52 weeks)
  The MG-ADL score is an 8-item patient-reported outcome (PRO) instrument. The MG-ADL targets symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The item responses are scored from 0 to 3, and the total score of MG-ADL is the sum of the 8 items and ranges from 0 to 24, with a higher score indicating more disability.
Change from Baseline in Quantitative Myasthenia Gravis (QMG) total score at the end of Week 6 of each TP | From Baseline to the end of Week 6 of each TP (up to 52 weeks)
  QMG score is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The QMG total score is obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3). The score ranges from 0 to 39, with lower scores indicating lower disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (10):
- Italy (3):
  - Mg0008 40290, Bologna
  - Mg0008 40144, Milan
  - Mg0008 40733, Napoli
- Japan (3):
  - Mg0008 20340, Fuchu-shi
  - Mg0008 20339, Ōbu
  - Mg0008 20343, Sagamihara
- Poland (2):
  - Mg0008 40734, Lodz
  - Mg0008 40155, Warsaw
- Taiwan (2):
  - Mg0008 20081, Taipei
  - Mg0008 20095, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org